CLINICAL TRIAL: NCT05012085
Title: Using Google Trends to Gauge the Popularity of Global Surgery Worldwide
Brief Title: Google Trends of Global Surgery
Status: Completed | Type: Observational
Sponsor: Association of Future African Neurosurgeons, Yaounde, Cameroon (Other)
Responsible Party: Sponsor
Other Study IDs: 0001
Record Dates: First submitted 2021-08-01; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Global Surgery; Global Health

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Investigation of Global Interest in Global Surgery — The investigators searched the terms "global surgery" and "global health" on Google Trends (Google Inc., CA, USA) from January 2004 to May 2021. The investigators identified time trends and compared the two search terms using SPSS v26 (IBM, WA, USA) to run summary descriptive analyses and Wilcoxon rank-sum tests.

SUMMARY:
Introduction Global surgery is a growing movement worldwide, but its expansion has not been quantified. Google Search is the most popular search engine worldwide, and Google Trends analyzes its queries to determine popularity trends. The investigators used Google Trends to analyze the regional and temporal popularity of global surgery (GS). Furthermore, the investigators compared GS with global health (GH) to understand if the two were correlated.

Methods The investigators searched the terms "global surgery" and "global health" on Google Trends (Google Inc., CA, USA) from January 2004 to May 2021. The investigators identified time trends and compared the two search terms using SPSS v26 (IBM, WA, USA) to run summary descriptive analyses and Wilcoxon rank-sum tests.

ELIGIBILITY:
Inclusion Criteria:

* Data point from Google Trends concerning Global Surgery
* Data point from Google Trends concerning Global Health
* Data point from Google Trends between January 2004 and May 2021

Exclusion Criteria:

* Data point from Google Trends before January 2004
* Data point from Google Trends after May 2021
* Data point from Google Trends outside the scope of Global Surgery or Global Health

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any data point included in the Google Trends database relevant to global surgery or global health.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Interest Levels | January 2004 to May 2021
  Level of interest in Global Surgery based on Google Trends

CONTACTS AND LOCATIONS:
Locations (1):
- Research Department, Association of Future African Neurosurgeons, Yaoundé, Cameroon